CLINICAL TRIAL: NCT02923102
Title: Effects of Recoverben® on Recovery After Exhaustive Exercise in Healthy People - a Randomized, Double-blind, Placebo-controlled Study With Parallel Design
Brief Title: Effects of Recoverben® on Recovery After Exhaustive Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vital Solutions GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BTS822/14
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers; Muscle Fatigue; Muscle Soreness
Keywords: Recovery; Muscle soreness; Lemon Verbena
MeSH Terms: conditions — Myalgia | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aloysia citriodora extract (Active Comparator): Dietary Supplement: Aloysia citriodora extract
  Interventions: Dietary Supplement: Aloysia citriodora extract
- Placebo Formulation (Placebo Comparator): Dietary Supplement: Maltodextrin (no active ingredient)
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Aloysia citriodora extract — 2 capsules with 200mg - daily dosage 400mg
  Other Names: Recoverben®
  Arms: Aloysia citriodora extract
Dietary Supplement: Maltodextrin — 2 capsules with 200mg - daily dosage 400mg
  Other Names: Placebo
  Arms: Placebo Formulation

SUMMARY:
The aim of the study is to investigate a pre and post workout supplementation (15 days) with Recoverben® , a Aloysia citriodora extract on recovery after exhaustive exercise. Effects will be investigated with 400mg Recoverben® and compared to placebo.

DETAILED DESCRIPTION:
The aim of the study is to investigate a pre and post workout supplementation (15 days) with Recoverben® , a Aloysia citriodora extract on recovery after exhaustive exercise. Effects will be investigated with 400mg Recoverben® and compared to placebo.

Targeted parameter will be determined at the beginning of the study and after supplementation, each. Parameter include maximal strength (MVC), muscle soreness (VAS), pain sensitivity (Algometry) and biomarkers (CK, IL-6, glutathione peroxidase).

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations
* Health volunteers: Subject is in good physical and mental health as established by medical his-tory, physical examination, electrocardiogram, vital signs, results of biochemistry and haematology
* Men and women
* Age ≥ 22 and ≤ 50 years
* BMI: 19-30 kg/m2
* Physically active 1-3 times per week
* Nonsmoker
* Able and willing to follow the study protocol procedures

Exclusion Criteria:

* Relevant history, presence of any medical disorder or chronic intake of medication/dietary supplements (e.g. polyphenols, anti-inflammatory or anti-oxidative drugs or supplements, antihyper-tensive drugs) potentially interfering with this study at screening.
* For this study clinically relevant abnormal laboratory, vital signs or physical findings at screening
* Diabetes or serious cardiovascular diseases
* Change of dietary habits within the 2 weeks prior to screening (for instance start of a diet high in vegetables and fruits (≥ 5 portions per day))
* Diet high in vegetables and fruits ≥ 5 portions per day
* Participants anticipating a change in their lifestyle or physical activity levels during the study.
* Subjects not willing to abstain from intake of analgesic medication (e.g. Aspirin) 24 hours prior to visit 2 until visit 5.
* Subjects with history of drug, alcohol or other substances abuse, or other factors limiting their ability to co-operate during the study.
* Known hypersensitivity to the study preparation or to single ingredients
* Pregnant subject or subject planning to become pregnant during the study; breast-
* Known HIV-infection
* Known acute or chronic hepatitis B and C infection
* Blood donation within 4 weeks prior to visit 1 or during the study.
* Subject involved in any clinical or food study within the preceding month

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Change of muscle soreness (VAS) over time | Chance over time after 10 days of supplementation (pre stress test and 3h, 24h, 48 h, 96h after stress test)
  In the current study, pain following eccentric exercise will be assessed by using a 100 mm visual analogue scale after the subjects performing a standardized movement.

SECONDARY OUTCOMES:
Monitoring of related adverse events | During study execution over 15 days
  Reporting of adverse effects to evaluate tolerability
Change of maximal concentric strength/ maximal voluntary contraction (MVC) over time | Chance over time after 10 days of supplementation (pre stress test and 3h, 24h and 48 h after stress test)
  Maximal concentric strength of the M. Quadriceps femoris will be assessed by measuring maximal isometric concentric strength using a dynamometer
Change of pressure pain (Algometry) over time | Chance over time after 10 days of supplementation (pre stress test and 3h, 24h and 48 h after stress test)
  The threshold for pressure induced pain will be measured using an algometer.
Change of retrospective pain (Likert scale) over time | Chance over time after 10 days of supplementation (pre stress test and 24h, 48h, 96h after stress test)
  Evaluation of the perceived pain retrospectively by using the Likert scale for muscle soreness
Change of creatine kinase over time | Chance over time after 10 days of supplementation (pre stress test and 3h, 24h and 48 h after stress test)
Change of of glutathione peroxidase over time | Chance over time after 10 days of supplementation (pre stress test and 24h and 48 h after stress test)
Change of interleukin-6 over time | Chance over time after 10 days of supplementation (pre stress test and 3h, 24h and 48 h after stress test)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Reule, Dr., Study Chair — BioTeSys GmbH
Locations (1):
- Biotesys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buchwald-Werner S, Naka I, Wilhelm M, Schutz E, Schoen C, Reule C. Effects of lemon verbena extract (Recoverben(R)) supplementation on muscle strength and recovery after exhaustive exercise: a randomized, placebo-controlled trial. J Int Soc Sports Nutr. 2018 Jan 23;15:5. doi: 10.1186/s12970-018-0208-0. eCollection 2018. PMID 29410606